CLINICAL TRIAL: NCT00545636
Title: The Influence of Education of Medical Team on Duration of Fasting Before Elective Medical Interventions Performed Under General Anesthesia in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unfortunately lacked manpower to carry out the study
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ze'ev Shenkman, MD, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: SHEBA-07-4879-ZS-CTIL
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Duration of Preoperative Fasting
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: education — The intervention is an education of the medical teams that instruct children to fast before the administration of general anesthesia

SUMMARY:
The purpose of the study is to examine if an education program of the medical teams can help implementation of of NPO (nothing-per-os)orders in children before anesthesia for ambulatory medical interventions under anesthesia and decrease unnecessary long fasting. We shall ask parents of such children to fill in a questionnaire regarding pre-anesthesia fasting and regular eating and drinking habits. Thereafter, all medical teams involved with the administration of NPO orders will receive an educational program to explain and implement the NPO orders as are recommended by the American Society of Anesthesiologists. We will examine if the educational program was successful in reducing unnecessary long period of fasting, and if such a program is not associated with increased rate of delay of cases.

ELIGIBILITY:
Inclusion Criteria:

* Children who are about to undergo anesthesia for elective medical interventions,
* Age 0-18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Education of the medical teams as to preoperative fasting time will aid in shortening of an unnecessary prolonged fasting | Immediate pre-anesthesia period (to assess lenth ofpreoperative fasting time)

CONTACTS AND LOCATIONS:
Overall Officials: Ze'ev Shenkman, MD, Principal Investigator — Sheba Medical Center, Department of Anesthsia C and Department of Anesthesia; Haim Berkenstadt, MD, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel